CLINICAL TRIAL: NCT05099705
Title: Testing a Family Service Navigator Program for Low-resourced Families of Young Children with Autism Spectrum Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Meghan Burke, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: University of Illinois
Record Dates: First submitted 2021-10-04; First posted 2021-10-29 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder; Mental Health Services
Keywords: Autism; Navigator; Services; Children; Low-resource
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Later in the project, a randomized controlled trial will be conducted. 40 participants will be in the intervention group and 15 participants will be in the non-personalized comparison group (i.e., information, training, and referral). Families will complete pre/post measures related to: intervention targets (except the ability to facilitate knowledge), service delivery outcomes, adaptive and maladaptive behavior, and autism symptoms. Information will also be collected via the treatment support system; such information will include the type and frequency of communication between the navigator and the family. Individual interviews will be collected with the navigator supervisor and the 20 navigators to identify barriers to the navigator model for low-resourced families.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Access to an FSN/TSS) (Experimental): 40 participants will be randomly assigned to the intervention group (i.e., to receive an FSN and have access to the TSS). The FSN may meet with the participant at least twice and provide navigation support.
  Interventions: Behavioral: Access to a Family Service Navigator and Treatment Support System
- Control Group (Access to Information, training and referral) (No Intervention): 15 participants will be randomly assigned to the non-personalized comparison group (i.e., information, training, and referral).

INTERVENTIONS:
Behavioral: Access to a Family Service Navigator and Treatment Support System — An RCT will be conducted. 40 participants will be randomly assigned to the intervention group and 15 participants to the non-personalized comparison group (i.e., information, training, and referral). The intervention group will have access to a navigator and the treatment support system.
  Arms: Intervention Group (Access to an FSN/TSS)

SUMMARY:
The purpose of this study is to develop and test a family navigator training and an app (a technology-based treatment support system) for low-resourced families of young children (aged 3-5) with autism. The hypothesis is that the navigator training and treatment support system will help enable navigators to support families of young children with autism in accessing needed services.

DETAILED DESCRIPTION:
The purpose of this project is to determine whether access to a family service navigator/treatment support system improves outcomes among families of young children (aged 3-5) from low-resourced communities. Pilot work includes interviews and pre/post surveys. Then, a randomized controlled trial will be conducted by randomly assigning families to navigators/treatment support systems or the non-personalized comparison condition (information, training, and referral services). Three-month, six-month, and nine-month follow-up survey data will be collected. Each of the 20 navigators will support two families. Intervention families will have access to the navigator and the treatment support system, which includes a dashboard showing their child's service needs, resources, and a platform to facilitate and document communication between navigators and families. The treatment support system will also allow the navigator supervisor to ensure fidelity of the navigators' support to the family. The statistician will randomize 55 families who meet the inclusionary criteria to each condition--40 individuals will receive navigator/treatment support system (intervention group) and 15 individuals will receive information, training, and referrals (comparison group).

ELIGIBILITY:
For the families in the clinical trial, there are the following inclusion and exclusion criteria:

Inclusion criteria:

* Be a parent who is in some way from a low-resourced community,
* Be the parent a child with autism between the ages of 3-5,
* Be age 18 or older,
* Want assistance with navigating service delivery systems,
* Be English speaking or Spanish-speaking,
* Be able to provide informed consent,
* Own a phone which can use the treatment support system (or be provided a phone from the Public Assistance Office or from the grant)

Exclusion criteria:

-Individuals who do not meet all inclusion criteria are by definition excluded.

For the navigators in the clinical trial, they must meet inclusion and exclusion criteria:

Inclusion Criteria:

* Agree to participate in the navigator training and become an navigator,
* Be a parent who is in some way from a low-resourced community,
* Be the parent a child with autism who is older than 5,
* Be age 18 or older, Be English speaking,
* Be able to provide informed consent,
* Own a phone which can use the treatment support system (or be provided a phone from the Public Assistance Office or from the grant)

Exclusion criteria:

-Individuals who do not meet all inclusion criteria are by definition excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge at 9 months | At the pre-survey and at the nine-month survey
  Called the Autism Knowledge Scale, a multi-item measure examining knowledge of autism services. There are 24 items with higher scores indicating more knowledge. Scale ranges from 0-24.
Change in Skills at 9 months | At the pre-survey and at the nine-month survey
  Called the Comfort with Advocacy Scale, A multi-item measure examining skills to identify, access, and receive services. There are 12 items with higher scores indicating greater advocacy. Scale ranges from 0 to 60.
Change in Advocacy at 9 months | At the pre-survey and at the nine-month survey
  Called the Advocacy Skills Scale, a multi-item measure examining the frequency of advocacy activities. There are nine items with higher scores indicating greater advocacy. Scale ranges from 9 to 45.
Change in Empowerment at 9 months | At the pre-survey and at the nine-month survey
  Called the Family Empowerment Scale, aa multi-item measure examining empowerment in family, services, and community/political environments. There are 34 items with higher scores indicating greater empowerment. Scale ranges from 0 to 136.
Change in Parenting self-efficacy at 9 months | At the pre-survey and at the nine-month survey
  Called the Self-Efficacy scale, a multi-item measure examining competence in parenting. There are nine items with higher scores indicating greater self-efficacy. Scale ranges from 0 to 36.
Change in Service Delivery Outcomes | At the pre-survey and at the three-month, six-month, and nine-month survey
  Called the adapted service measure scale, access to the type, number, and quality of services and unmet service needs. There are over 20 services with higher scores indicating needing greater services. Scale ranges from 0 to 20.
Change in Adaptive and maladaptive behavior at 9 months | At the pre-survey and at the nine-month survey
  Called the Vineland Adaptive Behavior Scale, a multi-item measure examining adaptive and maladaptive behavior. There are 100 items with higher scores indicating greater adaptive behavior. Scale ranges from 0 to 100.
Change in Social responsiveness at 9 months | At the pre-survey and at the nine-month survey
  Called the Social Responsiveness Scale, a multi-item measure to examine social responsiveness. There are sixty items with higher scores indicating greater social responsiveness. Scale ranges from 0 to 180.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Burke, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- University of Illinois at Urbana-Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data generated by this project will be an important part of the proposed activities of this research and will be carried out in several ways. All research resources developed in this project will be made readily available to the scientific community for non-profit research purposes. The main mechanism for the transfer of information will take the form of peer-reviewed publications and presentations/posters at scientific conferences. Information is collected from participants upon enrollment will be generated to a Global Unique Identifier. Annual reports with de-identified information will be presented to National Institute of Mental Health annually and more often upon request. By the completion of the project, all data will be de-identified and relevant documentation to facilitate data sharing will be available.
Supporting Information: Study Protocol
Time Frame: 7/2022-4/2025

REFERENCES:
- [Background] Magana, S., et al., Use of promotoras de salud in interventions with Latino families of children with IDD. International Review of Research in Developmental Disabilities, 2014. 47: p. 39-75
- [Background] Burke, M.M. and S.E. Goldman, Special education advocacy among culturally and linguistically diverse families Journal of Research in Special Educational Needs 2018. 1: p. 3-14.
- [Background] Maas, C.J. and J.P. Hox, Sufficient sample sizes for multilevel modeling. Methodology, 2005. 1: p. 86- 92.